CLINICAL TRIAL: NCT01364103
Title: Study About Predicting Fluid Responsiveness in Children Undergoing Neurosurgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, assistant professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: H-1012-118-345
Record Dates: First submitted 2011-05-24; First posted 2011-06-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Fluid Responsiveness
Keywords: pulse pressure variation; systolic pressure variation; central venous pressure; aortic blood flow velocity variation; pleth variability index

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Other: volume expansion — fluid loading of 10 mL/kg colloid (voluven)

SUMMARY:
The purpose of this study is to evaluate static and dynamic parameters, echocardiographic parameters, and pleth variability index for predicting fluid responsiveness in children. Children who need volume expansion will receive colloid 10 mL/kg. Blood pressure, heart rate, central venous pressure, systolic pressure variation, pulse pressure variation, delta down, aortic blood flow velocity variation, inferior vena cava diameter variation, and pleth variability index will be measure before and after volume expansion. Patients will be classified as responders to volume loading if stoke volume index increase by at least 15%.

ELIGIBILITY:
Inclusion Criteria:

* neurosurgery under general anesthesia
* < 8 years old

Exclusion Criteria:

* cardiac disease
* pulmonary, renal and hepatic disease
* infectious disease
* hematologic and muscular disease

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
stoke volume index | before and after volume loading (20 minutes)
  Volume loading will be performed for 20 minutes. Stroke volume will be meausred before and after volume expansion

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Derived] Byon HJ, Lim CW, Lee JH, Park YH, Kim HS, Kim CS, Kim JT. Prediction of fluid responsiveness in mechanically ventilated children undergoing neurosurgery. Br J Anaesth. 2013 Apr;110(4):586-91. doi: 10.1093/bja/aes467. Epub 2012 Dec 18. PMID 23250892